CLINICAL TRIAL: NCT05832255
Title: An Open-Label Investigation of the Effects of Sub-Perceptual Repeat Dosing of Psilocybin on the Behavioural and Cognitive Symptoms of Fragile X Syndrome in Adult Patients
Brief Title: An Investigation of Psilocybin on Behavioural and Cognitive Symptoms of Adults With Fragile X Syndrome
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Indefinite hold due to protocol revisions relating to the exclusion criteria for concurrent medications.
Sponsor: Nova Mentis Life Science Corp (Industry)
Collaborators: KGK Science Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22NMCFN01
Record Dates: First submitted 2023-03-08; First posted 2023-04-27 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Fragile X Syndrome; Behavior; Cognitive Dysfunction
Keywords: Fragile X Syndrome; Behavior; Cognitive Symptoms; Psilocybin; Microdose
MeSH Terms: conditions — Fragile X Syndrome; Behavior; Cognitive Dysfunction; Neurobehavioral Manifestations | interventions — Psilocybin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Psilocybin, 1.5 mg (Experimental): Participants will take one capsule containing 1.5 mg psilocybin with a glass of water every other day for a period of 28 days. Dosing schedule will be same for all participants with the drug taken at days 1, 3, 5, 7, 9, 11, 13, 15, 17, 19, 21, 23, 25, 27, and no treatment taken on alternating days. No subject shall be provided with more than five capsules (7.5mg psilocybin) at any one time to prevent diversion to the illicit market. If a dose is missed, participants are instructed to skip that dose and continue with their regularly scheduled medications. Participants are not to take >1 capsule per day.
  Interventions: Drug: Psilocybin, 1.5 mg

INTERVENTIONS:
Drug: Psilocybin, 1.5 mg — Blister packs will contain five capsules of the study drug, Psilocybin 1.5mg. Subjects will be given blister packs with weekly doses at each visit including baseline (day 1), day 8, day 15, day 21, and day 28. Weekly blister packs will contain five doses (1-2 extra capsules depending on the week) to accommodate for flexibility in scheduling. Unused and open packages will be returned to study staff at each visit after baseline.

SUMMARY:
Diverse symptomatology makes Fragile X Syndrome (FXS) difficult to treat, and currently there are no approved prevention or treatment methods for FXS. Current therapies, including pharmaceutical and behavioural interventions, offer a patchwork of solutions that have limited efficacy and high toxicity. The current study aims to examine psilocybin as a safe treatment alternative with the ability to improve markers of cognition, communication, mood, behavior as well as markers of neuroinflammation, serotonin levels in exosomes, and neuroplasticity at sub-hallucinogenic doses (microdosing).

The overall objective of this study is to assess the feasibility of low-dose psilocybin as a therapeutic option for individuals living with FXS and to improve diagnostic parameters of FXS, as well as therapeutic responses with the use of biomarkers.

DETAILED DESCRIPTION:
A total of 10 subjects who meet all the inclusion criteria and does not meet any of the exclusion criteria will be enrolled into the study. Any subjects prematurely terminated from the study will be replaced to ensure 10 subjects complete the study. A study coordinator will contact referring clinicians, caregivers, and subjects to pre-screen for initial eligibility. Those deemed eligible will be invited for an in-person screening along with the participating caregiver. The screening visit will be approximately two hours long and will consist of informed consent, diagnostic interview, physical examination, drugs of abuse test (DOA), ECG, medical/treatment history review, and demographic forms. A pregnancy test will be performed on females of child-bearing during screening, baseline, and end-of-study visits. All eligible subjects will enter the treatment arm of the study.

Subjects and caregivers will return to the clinic for a baseline visit within three weeks of their screening completion. Baseline visit will include saliva/buccal swab collection, and clinician and self-report assessments for subjects and caregivers. These assessments will include the Vineland Adaptive Behavior Scales-Third Edition (VABS-3), Clinical Global Impressions-Improvement scale (CGI-I), Visual Analog Scale-Treatment Satisfaction (VAS-TS), the Anxiety, Depression and Mood Scale (ADAMS), and the Systematic Assessment For Treatment Emergent Events (SAFTEE). Digital assessments may also be performed at the baseline visit or at home at the discretion of the qualified investigator. Digital assessments will include the NIH Toolbox Cognitive Battery Modified for Intellectual Disabilities (NIH-TCB), the Trail Making Test (TMT), and the Multifaceted Empathy Test (MET).

The study drug will be dispensed in blister packs to monitor adherence and improve subject compliance. Blister packs will be prepared and distributed at each subsequent visit. Subjects will return to the clinic for study visits on day 8, 15, 22, and 28 (study end date). Subjects and caregivers will complete the assessments described above. Subjects will provide additional saliva/buccal swab samples at day 15 and day 28.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 50 years of age
2. BMI > 18.3
3. Diagnosis of Fragile X syndrome with a molecular genetic confirmation of the full FMR1 mutation (>200 CGG repeats) or the other loss of function mutations of the FMR1 gene (SNVs and deletions of the gene) based on evidence provided by caregiver from prior assessment
4. IQ between 40 and 85 points as reported by caregiver based on prior assessment
5. Subject has the ability to understand and provides voluntary, written, informed consent to participate in the study

   Or,

   For subjects who are not their own legal guardian, or do not have the capacity to provide informed consent, subject's parent/legal authorized guardian is able to understand and sign an informed consent form to participate in the study.
6. Caregiver (parent, guardian, or other legally authorized representative) who is willing to participate in the whole study and provides informed consent
7. Subject is able to swallow tablets and capsules
8. Individual is not of child-bearing potential, defined as those who have undergone a sterilization procedure (e.g. hysterectomy, bilateral oophorectomy, bilateral tubal ligation, complete endometrial ablation) or have been post-menopausal for at least 1 year prior to screening

Or,

Individuals of child-bearing potential must have a negative baseline urine pregnancy test and agree to use a medically approved method of birth control for the duration of the study. All hormonal birth control must have been in use for a minimum of three months. Acceptable methods of birth control include:

* Abstinence (only in cases when abstinence is the usual and customary form of birth control for the participant)
* Hormonal contraceptives including oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (Depo-Provera, Lunelle), or hormone implant (Norplant System)
* Double-barrier method
* Intrauterine devices
* Non-heterosexual lifestyle or agrees to use contraception if planning on changing to heterosexual partner(s)
* Vasectomy of partner at least 6 months prior to screening

Exclusion Criteria:

1. Individuals who are pregnant, breast feeding, or planning to become pregnant during the study
2. Allergy, sensitivity, or intolerance to the investigational product's active or inactive ingredients
3. Regular use of medications that may have problematic interactions with psilocybin, including but not limited to dopamine agonists, MAO inhibitors, N-methyl-D-aspartate (NMDAR) antagonists, antipsychotics, and stimulants
4. Urine drug test containing non-prescribed drugs of abuse (non-prescribed opioids, benzodiazepines, amphetamines, phencyclidine, cocaine) at screening and day of first treatment. Urine cannabinoid concentrations >50 ng/ml will suggest heavy marijuana use and will be a threshold for excluding potential subjects
5. Having uncontrolled hypertension defined as an average systolic blood pressure ≥140 mmHg or an average diastolic blood pressure ≥90 mmHg, with at least 4 BP assessments completed.
6. Have any of the following cardiovascular conditions: coronary artery disease, congenital long QT (time from the start of the Q wave to the end of the T wave) syndrome, cardiac hypertrophy, cardiac ischemia, congestive heart failure, myocardial infarction, tachycardia, artificial heart valve, a clinically significant screening ECG abnormality, or any other significant cardiovascular condition
7. Significant cardiovascular event in the past 6 months. Participants with no significant cardiovascular event on stable medication may be included after assessment by the QI on a case-by-case basis
8. Subjects with a history of seizure disorder except those who are currently receiving treatment with anti-epileptics and have been seizure-free for 3 months preceding screening or have been seizure-free for 3 years if not currently receiving anti-epileptics.
9. Reported history of moderate to severe hepatic impairment
10. Type I or insulin-dependent Type II diabetes
11. Meet DSM-5 criteria for schizophrenia spectrum or other psychotic disorders, including major depressive disorder with psychotic features, or Bipolar I or Bipolar II Disorder
12. Meet DSM-5 criteria for a moderate or severe alcohol or drug use disorder in the past 12 months
13. Subjects who plan to initiate or change pharmacologic or non-pharmacologic interventions during the course of the study
14. Medical illness based on physical examination, ECG and routine testing that may complicate cardiovascular safety or drug metabolism or excretion, such as metabolic disease, severe cardiac disease, or kidney or liver failure as assessed by the QI. QI assessments will be based on clinical history provided by caregivers and/or physicians. Any participant requiring further assessment will be referred accordingly or excluded by the QI on a case-by-case basis.*
15. Current or history of any significant diseases of the gastrointestinal tract, exceptions to be determined by the QI
16. Unstable hypertension. Treatment on a stable dose of medication for at least 3 months will be considered by the QI on a case-by-case basis
17. Major surgery in the past 3 months or individuals who have planned surgery during the course of the study. Participants with minor surgery will be considered on a case-by-case basis by the QI
18. Participation in other clinical research studies 30 days prior to enrollment as assessed by the QI.
19. Any other condition or lifestyle factor, that, in the opinion of the QI, may adversely affect the participant's ability to complete the study or its measures or pose significant risk to the participant * Blood draw to obtain laboratory samples for analysis will be avoided in this study due to the undue stress it places on this clinical population and the high safety profile of the medication at the dosage being used.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-03-28 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Retention rate associated with 10 participants progressing to study completion. | baseline to day 28
  Study completion is defined as completing the 28-day treatment period and the final in-clinic study visit.
Compliance with study dosing regimen as measured by the Visual Analogue Scale for Dosing (VAS-D). | baseline to day 28
  Participants will be monitored for compliance using electronic compliance checks via the remote patient reported outcomes system through recording consumption in the treatment diary. Participants and caregivers will receive daily notifications via their preferred format (i.e., email, text) during agreed upon dosage windows. Notification will include a reminder to complete a post-dosage Visual Analogue Scale for Dosing (VAS-D) to monitor for any side effects which can be submitted electronically. Failure to complete the VAS-D within the day of dosing will trigger a call from study personnel to the participant in order to do a compliance check. Study personnel will note any deviations and all points of contact with participants regarding compliance checks.
Compliance with study dosing regimen as measured by the quantity of unused investigational product returned to the study clinic. | baseline to day 28
Adherence with completion of diaries monitoring participant and caregiver reported outcomes. | baseline to day 28
  Adherence with study requirements for patient reported and caregiver reported outcomes (i.e., diaries) will be monitored using a remote patient reported outcomes system. Adherence will be assessed by determining the number of completed patient/caregiver diaries divided by the number of diaries expected to be completed.
Adherence with completion of questionnaires monitoring participant and caregiver reported outcomes. | baseline to day 28
  Adherence with study requirements for patient reported and caregiver reported outcomes (i.e., questionnaires) will be monitored using a remote patient reported outcomes system. Adherence will be assessed by determining the number of completed patient/caregiver questionnaires divided by the number of questionnaires expected to be completed.
The number of late entries for diaries monitoring patient reported and caregiver reported outcomes. | baseline to day 28
The number of late entries for questionnaires monitoring patient reported and caregiver reported outcomes. | baseline to day 28
Satisfaction with study questionnaire. | baseline to day 28

SECONDARY OUTCOMES:
Change from baseline in standardized measures of behavioral rigidity using the ratings of repetitive and stereotyped behaviors from the revised Repetitive Behavior Scale (RBS-R). | baseline, day 15, day 28
Change in standardized measures of empathy using the communication domain of the Vineland Adaptive Behavior Scales- Third Edition (VABS-3). | baseline, day 15, day 28
Change in standardized measures of empathy using the overall score on the Multifaceted Empathy Test (MET). | baseline, day 15, day 28
Change in standardized measures of expressive and receptive language skills using the communication domain of the Vineland Adaptive Behavior Scales- Third Edition (VABS-3). | baseline, day 15, day 28
Change in standardized measures of expressive and receptive language skills using the overall score on the Multifaceted Empathy Test (MET). | baseline, day 15, day 28
Changes in standardized measures of behavioral symptoms as measured by the Aberrant Behavior Checklist (ABC) with particular focus on ratings of repetitive/ritualistic behaviors from baseline to end of study. | baseline, day 8, day 15, day 21, day 28
Changes in standardized measures of behavioral symptoms as measured by the Aberrant Behavior Checklist (ABC) with particular focus on ratings of aggressive behaviors from baseline to end of study. | baseline, day 8, day 15, day 21, day 28
Changes in standardized measures of behavioral symptoms as measured by the revised Repetitive Behavior Scale (RBS-R) with particular focus on ratings of repetitive/ritualistic behaviors from baseline to end of study. | baseline, day 8, day 15, day 21, day 28
Changes in standardized measures of behavioral symptoms as measured by the revised Repetitive Behavior Scale (RBS-R) with particular focus on ratings of aggressive behaviors from baseline to end of study. | baseline, day 8, day 15, day 21, day 28
Changes in standardized measures of behavioral symptoms as measured by the Clinical Global Impressions (CGI) scale with particular focus on ratings of repetitive/ritualistic behaviors from baseline to end of study. | baseline, day 8, day 15, day 21, day 28
Changes in standardized measures of behavioral symptoms as measured by the Clinical Global Impressions (CGI) scale with particular focus on ratings of aggressive behaviors from baseline to end of study. | baseline, day 8, day 15, day 21, day 28
Changes in standardized measures of behavioral symptoms with particular focus on ratings of aggressive behaviors from baseline to end of study. | baseline, day 8, day 15, day 21, day 28
  Changes in behavioral symptoms will be measured via the Aberrant Behavior Checklist (ABC), revised Repetitive Behavior Scale (RBS-R), and Clinical Global Impressions (CGI) scale.
Changes in overall cognition scores as measured by the NIH Toolbox Cognitive Battery Modified for Intellectual Disabilities (NIH-TCB). | baseline, day 28
Changes in overall cognition scores as measured by the Trail Making Test (TMT)-digital version. | baseline, day 28
Changes in overall cognition scores as measured by the Behavior Rating Inventory of Executive Function-Adult Version (BRIEF-A). | baseline, day 28
Changes in standardized measures of cognitive flexibility as measured by the NIH Toolbox Cognitive Battery Modified for Intellectual Disabilities (NIH-TCB) from baseline to end of study. | baseline, day 28
Changes in standardized measures of cognitive flexibility as measured by the Trail Making Test (TMT)-digital version from baseline to end of study. | baseline, day 28
Changes in standardized measures of cognitive flexibility as measured by the Behavior Rating Inventory of Executive Function-Adult Version (BRIEF-A) from baseline to end of study. | baseline, day 28
Changes in standardized measures of anxiety and depression with corresponding changes in ratings of overall wellbeing. | baseline, day 8, day 15, day 21, day 28
  Changes in anxiety, depression, and overall wellbeing will be measured via the Anxiety, Depression and Mood Scale (ADAMS).

OTHER OUTCOMES:
To improve diagnostic phenotyping of FXS through analysis of biomarkers using buccal swab and saliva samples. | baseline, day 15, day 28
  Machine learning algorithms will be applied to analyze and establish clustering and/or correlation between diverse datasets to help stratify adults with FSX according to subtle differences in mRNA neuroinflammatory biomarkers, serotonin signaling, and behavior.
To characterize the role of psilocybin as a modulator of neuroinflammation through analysis of mRNA neuroinflammatory biomarkers using saliva samples from baseline to study end. | baseline, day 15, day 28
  mRNA analysis will include a panel with 52 genes including cytokines, cytokine targets, neurotransmission, serotonin signaling, membrane channel, DNA damage repair, and growth factors.
To characterize the role of psilocybin as a modulator of neuroinflammation through analysis of mRNA neuroinflammatory biomarkers using buccal swabs from baseline to study end. | baseline, day 15, day 28
  mRNA analysis will include a panel with 52 genes including cytokines, cytokine targets, neurotransmission, serotonin signaling, membrane channel, DNA damage repair, and growth factors.
To characterize the role of psilocybin as a modulator of neuroinflammation through analysis of serotonin levels using saliva samples from baseline to study end. | baseline, day 15, day 28
To characterize the role of psilocybin as a modulator of neuroinflammation through analysis of serotonin levels using buccal swabs from baseline to study end. | baseline, day 15, day 28
The incidence of pre-emergent and post-emergent adverse events. | baseline to 28 days
The incidence of clinically significant changes in blood pressure (BP). | baseline, day 8, day 15, day 21, day 28
The incidence of clinically significant changes in heart rate (HR). | baseline, day 8, day 15, day 21, day 28

CONTACTS AND LOCATIONS:
Overall Officials: David Crowley, MD, Principal Investigator — KGK Science Inc.; Marvin Hausman, MD, Study Chair — Nova Mentis Life Science Corp
Locations (1):
- KGK Science Inc., London, Ontario, Canada